CLINICAL TRIAL: NCT00726466
Title: A Phase I Study of the Inhibition of LFA-1 to Intercellular Adhesion Molecule-1 (ICAM-1) Using Subcutaneous Efalizumab Combined With Intravitreal Ranibizumab in the Treatment of Age-Related Macular Degeneration (SEIRA)
Brief Title: Study of Efalizumab Combined With Intravitreal Ranibizumab in the Treatment of Age-Related Macular Degeneration
Acronym: SEIRA
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Vitreous -Retina- Macula Consultants of New York (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Jason S. Slakter, MD, Vitreous Retina Macula Consultants of New York
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF4385s
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Age Related Macular Degeneration; AMD; CNV
Keywords: Age Related Macular Degeneration; AMD; CNV
MeSH Terms: conditions — Macular Degeneration | interventions — efalizumab; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): This is an open-label, study of 0.5 mg intravitreal dose of Ranibizumab in combination with 1 mg/kg/wk subcutaneous dose of Efalizumab in in subjects with AMD.
  Interventions: Drug: Efalizumab, Ranibizumab

INTERVENTIONS:
Drug: Efalizumab, Ranibizumab

SUMMARY:
Efalizumab is an immunosuppressive recombinant humanized IgG1 monocolonal antibody (150 Kd) that binds to human CD11a (1) and is used for the treatment of plaque psoriasis. Efalizumab was derived from the humanization of the murine efalizuman monoclonal antibody MHM24, which recognizes human and chimpanzee CD11a. Humanization of MHM24 was accomplished by grafting the murine complementarity determining regions (hypervariable region) into consensus human IgG1/ heavy and light chain sequences (Werther et al 1996). These same consensus human immunoglobulin sequences have been successfully used in the humanization of other murine antibodies, including those targeted to HER2 and IgE. Efalizumab inhibits the binding of LFA-1 to intercellular adhesion molecule-1 (ICAM-1) thereby inhibiting the adhesion of leukocytes to other cell types.

Ranibizumab is a recombinant, humanized, Fab fragment of a mouse monoclonal antibody targeted against VEGF. As VEGF binds to cellular receptors, it stimulates angiogenesis and vascular leakage. Blockade of VEGF by ranibizumab leads to reduced stimulation of cell proliferation and permeability resulting in inhibition of angiogenesis and decreased leakage. Ranibizumab intravitreal administration in neovascular AMD patients has been shown to effectively reduce vascular leakage and growth of CNV and to stabilize or improve visual function.

To further improve visual acuity, a combination therapy using efalizumab and ranibizumab is proposed. Efalizumab could target the adhesion factors that precede angiogenesis and improve the outcome for AMD patients in combination with the anti-VEGF agent, Ranibizumab.

DETAILED DESCRIPTION:
This is an open-label, study of 0.5 mg intravitreal dose of Ranibizumab in combination with 1 mg/kg/wk subcutaneous dose of Efalizumab in in subjects with AMD. 10 subjects from 1 site will be enrolled in this study. Subject accrual into the trial is expected to be completed within 6 months.

All subjects will be evaluated monthly with a full ocular examination, visual acuity measurement (ETDRS chart at distance of 4 meters), OCT, and adverse event monitoring. Fluorescein Angiography (FA) and fundus photos will be done at BSL, Months 3, 6, 9 and 12.

Subjects will receive efalizumab 1mg/kg weekly subcutaneous injections for 24 weeks. Subcutaneous Efalizumab injections can be self administered after an initial teaching session in office on Day 0.

Subjects will receive six initial doses of 0.5 mg/eye intravitreous monthly injections of ranibizumab (Day 0, Months 1, 2, 3, 4 and 5) with scheduled follow-up visits monthly for 12 months. Re-treatment after the first six injections will be on an as-needed basis, based on predefined criteria.

3.2 RATIONALE FOR STUDY DESIGN

The rationale for the study is as follows:

* Phase III studies of patients with primary or recurrent choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD) treated with repeated intravitreal injections of 0.5 mg of ranibizumab showed evidence for bioactivity, safety, and tolerability (Rosenfeld 2006);
* Phase III studies of patients with chronic moderate to severe plaque psoriasis treated with weekly subcutaneous efalizumab injections of 1mg/kg showed evidence for bioactivity, safety, and tolerability (Dubertret 2006);
* A Phase I study of patients with uveitis treated with subcutaneous efalizumab injections of 1mg/kg in patients with uveitic macular edema is currently enrolling (ClinicalTrials.gov Identifier: NCT00280826)
* Combination therapy of an iCAM-1 inhibitor and an anti-VEGF agent may offer increased treatment benefit in the management of age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Demonstrate understanding of and ability to perform weekly self sub-cutaneous injections.
* Subjects of either gender, Age > 50 years
* Best corrected visual acuity in the study eye between 20/40 and 20/320.
* Subfoveal choroidal neovascularization, secondary to age related macular degeneration. 6-10 anti-VEGF treatments allowed prior to enrollment.
* Presence of subretinal fluid and/or cystoid retinal edema on OCT.
* Presence of fibrosis, hemorrhage, serous pigment epithelial detachments, tear (rip) of the retinal pigment epithelium or other hypofluorescent lesions should not obscure greater than 50% of the CNV lesion.
* Annual immunization completed at least 4-6 weeks prior to BSL.
* Clear ocular media and adequate papillary dilation to permit good quality stereoscopic fundus photography
* Ability to return for all study visits

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactation.
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Had prior treatment with Photodynamic Therapy (PDT).
* Had treatment with anti-VEGF agents within 30 days prior to BSL.
* Had treatment with Kenalog within 6 months prior to BSL.
* Had treatment with Dexamethaosne within 30 days prior to BSL.
* Had ocular surgery within the past 60 days in the study eye.
* Concurrent use of more than two therapies for glaucoma.
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure >30 mm Hg despite treatment with anti-glaucoma medication).
* Concurrent use of systemic anti-VEGF agents
* Has active infection in the study eye.
* Inability to obtain photographs to document CNV.
* Has received investigational therapy within 60 days prior to study entry.
* Patients with significantly compromised visual acuity in the study eye due to concomitant ocular conditions.
* Have a history of hypersensitivity to efalizumab or any of its components
* Current or history of prior treatment of psoriasis with subcutaneous efalizumab within 6 months of study entry.
* Have a history of ongoing uncontrolled serious bacterial, viral, fungal, or atypical mycobacterial infection. This includes diagnoses that required more than 2 weeks of therapy, such as endocarditis and osteomyelitis, which have been treated in the past 6 months. In addition, if the subject is currently receiving antibiotics, antivirals, or antifungals for an infection or for suppression or prophylaxis for any diagnosis.
* Have a history of opportunistic infections (e.g. systemic fungal infections, parasites)
* Have the presence or history of malignancy, including lymphoproliferative disorders. Subjects with a history of fully resolved basal or squamous cell skin cancer may be enrolled.
* Have a history of thrombocytopenia, clinically significant hemolytic anemia, or unexplained anemia.
* Have a platelet count < 100,000 cells/uL
* Has other conditions the investigator considers to be sound reasons for exclusion (e.g., lack of motivation, history of poor compliance, concomitant illnesses, personality disorder, mental condition, drug abuse, use of neuroleptics, physical or social condition predicting difficulty in long-term follow-up).
* Patients receiving immunosuppressive agents (including but not limited to cyclosporine, methotrexate, azathioprine, mycophenolate mofetil and systemic steroids) are excluded from the screening visit until study completion
* All acellular, live and live-attenuated vaccines are excluded from 14 days prior to the first dose of efalizumab until a minimum of 4 weeks after the last dose of efalizumab
* Has an allergy to sodium fluorescein dye.
* Inability to comply with study or follow-up procedures.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03

PRIMARY OUTCOMES:
• Safety and tolerability of 0.5 mg intravitreal dose of Ranibizumab in combination with 1 mg/kg/wk subcutaneous dose of Efalizumab in the treatment of age-related macular degeneration using the incidence and severity of adverse events through Month 6.

SECONDARY OUTCOMES:
The secondary outcomes of this study are as follows: • Mean change in ETDRS BCVA at Months 6 and 12. • Mean change in central retinal thickness per OCT at Months 6 and 12 • Mean change in lesion and CNV size as determined by FA at Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Jason S Slakter, MD, Principal Investigator — Vitreous -Retina- Macula Consultants of New York
Locations (1):
- Vitreous Retina Macula Consultants of New York, New York, New York, United States

REFERENCES:
- See also: Study site — http://www.vrmny.com